CLINICAL TRIAL: NCT05283213
Title: Elaboration d'un Score Clinico-biologique Innovant Pour la détection précoce de l'Insuffisance rénale aiguë associée à la chirurDevelopment of an Innovative Clinico-biological Score for the Early Detection of Acute Renal Failure Associated With Cardiac Surgery. Gie Cardiaque. Monocentric Prospective Study
Brief Title: Development of an Innovative Clinico-biological Score for the Early Detection of Acute Renal Failure Associated With Cardiac Surgery.
Acronym: DETECT-AKI
Status: Completed | Type: Observational
Sponsor: Nantes University Hospital (Other)
Collaborators: Roche Pharma AG (Industry); ThermoFisher Scientific Brahms Biomarkers France (Industry)
Responsible Party: Sponsor
Other Study IDs: RC22_0108
Record Dates: First submitted 2022-02-23; First posted 2022-03-16 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2026-01

CONDITIONS: Acute Kidney Injury
Keywords: AKI, extracorporal circulation, nephroprotection
MeSH Terms: conditions — Acute Kidney Injury

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Months
Biospecimen Retention: Samples With DNA — whole blood and urine
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Early biomarkers of acute kidney injury — The biomarkers tested will be:
  * creatinine levels [pre-, post-CC, H6],
  * Plasma NGAL [Pre-, Post-CC, H6].
  * Urinary NGAL [H6]
  * Plasma cystatin C [Pre-CC, Post-CEC & H6],
  * plasma HI [pre-, post-CC, H6],
  * plasma IL-6 [post-CC, H6],
  * uremia [pre-, post-CC, H6],
  * urinary DKK3 [pre-CC],
  * urinary CCL-14 [H6],
  * plasma angiopoietin-2 [H6],
  * plasma PENK-A [H6]
  These biomarkers will, if necessary, be corrected for hemodilution or dilution of urine, if any, using [pre-, post-CC, H6] protein and [pre-, post-CC, H6] creatinine, respectively.

SUMMARY:
The prediction and early detection of acute renal failure associated with cardiac surgery (ARF-CS) are desirable in order to try to reduce its magnitude. Indeed, its incidence is high (29 to 36%, reaching up to 81% in some series, depending on the vulnerability of the target population) and its consequences are often serious: prolongation of the length of stay in the intensive care unit and in hospital, death, and evolution towards chronic renal failure, possibly end-stage (justifying long-term extra-renal purification and/or renal transplantation). The challenge is all the more crucial given the high volume of cardiac surgery. In this context, the objective of identifying early on patients at high risk of developing AKI-CC - and therefore eligible for "nephroprotective" measures has generated, in the last decade, a strong interrest around preoperative scores and biomarkers. Thus, more than ten models predicting AKI-CC have been developed and more than 150 candidate biomarkers have been identified since 2004. This insterest is not waning. The DETECT-AKI project aims to evaluate, in a large population (N=400 patients) with varied patient profiles, not only the performance of the most innovative and promising preoperative scores and biomarkers described in the literature, but also the combination of biomarkers with relevant perioperative clinical and biological data in the framework of a clinico-biological score for the early identification of AKI-CC

DETAILED DESCRIPTION:
The DETECT-AKI study aims at establishing an innovative composite score, the basis for decision making in the early initiation of nephroprotection measures. This score will include early clinical and biological data before, during and after surgery and may therefore include one or more modern biomarkers. The DETECT-AKI study foresees from the outset the internal validation of the score by bootstrap method: first essential step for the subsequent application of the established score. This is also one of the strengths of the study.

ELIGIBILITY:
Inclusion Criteria:

* Adults undergoing scheduled, combined, cardiac surgery with CEC.
* "Combined" cardiac surgery (as opposed to simple cardiac surgery, which is less likely to result in ARF-CC) involves:

  * 2 heart valves (and possibly other procedures) or ≥2 types of procedures among coronary artery bypass graft(s), valve, myocardial, and thoracic aortic surgery.
* A "scheduled" surgical procedure implies that the patient was added to the operative schedule more than 24 hours before the procedure.

Exclusion Criteria:

* unscheduled cardiac surgery
* at least one session of extra-renal purification in the week prior to surgery
* Patient refusal to participate in this research,
* participation in a study with a possible impact on the incidence of AKI-CC
* pregnant woman
* minor, adult under guardianship, protected person.
* no biomarker concentrations were measured and no clinico-biological scores were determined,
* no pre-CEC creatinine assay is available,
* the patient dies before H48 unless AKI-CC has occurred in the interim,
* the patient withdraws consent to participate in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults undergoing scheduled, combined, cardiac surgery with CC inducing possible acute kidney injury as a consequence
Sampling Method: Non-Probability Sample
Enrollment: 400 (Actual)
Dates: Start 2022-11-22 (Actual); Primary Completion 2025-03-10 (Actual); Study Completion 2025-03-10 (Actual)

PRIMARY OUTCOMES:
composite score | From pre-CC to 6th hour post CC
  The primary endpoint will be ASCroc associated with the DETECT-AKI composite score established at H6.
  AKI-CC will be based on the current international definition (elevation of creatinine and/or occurrence of oliguria within 48 h postoperatively). Internal validation of the score will be based on a bootstrap resampling method.

SECONDARY OUTCOMES:
Early renal biomarkers performance (creatininemia, urinary TIMP*IGFBP7, plasma and urinary NGAL, plasma Cystatin C / Plasma Hemolysis Index (PH) / interleukin-6, uremia and urinary DKK3) | From pre-CC to 6th hour post CC
  Comparison of individual biomarker performance in identifying AKI-CC (all stages) at or before the 6th hour post-CC. The performance of an isolated measurement (at a given perioperative time) of a given biomarker will be analyzed, as well as the variation over time of the concentration of this biomarker (diagnostic performance of the biomarker kinetics).
Score performance of early renal biomarkers (creatininemia, urinary CCL-14, plasma and urinary NGAL, plasma Cystatin C, IH, IL6, angiopoietin-2, PENK-A, uremia and urinary DKK3) | From pre-CC to 6th hour post CC
  Comparison of the performance of scores proposed in the literature for the prediction of AKI-CC (all stages) on pre-operative data:
  * Cleveland Clinic Foundation score (dialysis risk for severe AKI (grade III) after cardiac surgery from 0 to 13 (highest risk)
  * Mehta score (calculator that estimates the risk of dialysis after cardiac surgery on demographic and antecedent data for severe AKI (grade III)
  * Ng score (same as Metha score without endocarditis data)
  * Simplified Predictive Index (for renal replacement therapy (RRT) after cardiac surgery from 0 to 8 (highest risk)
  * Leicester score (predicts CSA-AKI of any stage after cardiac surgery using a formula taking into account KDIGO stage but without diuresis)
  * EuroSCORE II (calculator that estimates the risk of dialysis after cardiac surgery on demographic, antecedent data using a formula)
Score and biomarkers performance for prediction | From pre-CC to 6th hour post CC
  Comparison of the individual performances of scores and biomarkers for the prediction or early detection of moderate to severe AKI-CC (KDIGO stages II and III), rather than AKI-CC of any stage.
Algorithm | From pre-CC to 6th hour post CC
  Construction of a triage algorithm for early classification of patients according to risk of developing AKI-CC (any stage) with pre-operative data as well as per-operative and early post-operative data
Biomarkers performance in AKI persistance (creatininemia, urinary TIMP*IGFBP7, plasma and urinary NGAL, plasma Cystatin C / Plasma Hemolysis Index (PH) / interleukin-6, uremia and urinary DKK3) | beyond 48th hour post CC to 7 days
  Evaluation of the performance of biomarkers to predict the transient or persistent nature of AKI-CC beyond the 48th hour in patients who have developed AKI-CC.
Sensitivity analysis | At 7th days
  Sensitivity analysis: analysis of the performance of the composite score using
  * the strict KDIGO definition of AKI-CC, i.e. setting the observation time for the criterion "relative rise in creatinine" at 7 days.
  * omitting the diuresis criterion from the definition, as diuresis is sometimes considered misleading in the context of cardiac surgery (due to the frequent use of diuretics, for example).

CONTACTS AND LOCATIONS:
Overall Officials: Karim Lakhal, MD, Principal Investigator — Nantes UH
Locations (1):
- Nantes UH, Nantes, France

IPD SHARING:
Plan to Share IPD: No